CLINICAL TRIAL: NCT03577652
Title: The Optimal Strategy of Switching From Clopidogrel to Ticagrelor in Patients With Complexity of Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, General Hospital of Shenyang Military Region, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180621
Record Dates: First submitted 2018-06-20; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease; Ticagrelor
Keywords: Ticagrelor; Clopidogrel; Switching strategy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ticagrelor, 90mg, 12h (Experimental)
  Interventions: Drug: Ticagrelor
- Ticagrelor, 90mg, 24h (Experimental)
  Interventions: Drug: Ticagrelor
- Ticagrelor, 180mg, 24h (Experimental)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor, 90mg, 90mg twice daily

SUMMARY:
The study is to further exploring the optimal switching strategy by evaluating the pharmacodynamic responses as well as adverse events in patients with complexity of coronary artery disease managed by percutaneous coronary intervention (PCI). All participants will be divided into three groups and recieving ticagrelor 90mg plus aspirin 100mg at 12 hours after the last dose of clopidogrel; recieving ticagrelor 90mg plus aspirin 100mg at 24 hours after the last dose of clopidogrel; recieving ticagrelor 180mg plus aspirin 100mg at 24 hours after the last dose of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75
2. Patients with complexity of CAD determined by coronary angiography and implanted stent successfully
3. Taking clopidogrel 75mg daily over 5 days or paients never took clopidogrel previously should receive 300-600mg drugs at least 12 hours before coronary angiography
4. Agreeing to participate in this trial and signed the written informed consent.

Exclusion Criteria:

1. They contraindicated with ticagrelor (including: allergying to ticagrelor or its active metabolite
2. Concomitanting therapy with a strong cytochrome P-450 3A inhibitor or inducer
3. Previous intracranial haemorrhage or ongoing bleeds
4. Moderate or severe hepatic impairment)
5. Having a previous medication with ticagrelor or long term anticoagulation
6. Having a history of asthma or chronic obstructive pulmonary disease (COPD) and recurrent attacked
7. Having an uncontrolled hypertension>180/110mmHg
8. Having a hemoglobin<100g/L 9.Having a platelet counts<100×10^9/L
9. Having severe renal impairment (clearance<30mL/min)
10. Having a history of hepaein-induced thrombocytopenia (HIT)
11. Having a pregnancy or were during lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Platelet function assessments | 7 Days
  The primary endpoint was the comparations between the three projects for the value changes of maximal platelet aggregation (MPA) measured by Light Transmittance Aggregometry (LTA) at 2 hours after switching strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Yao Y, Wang P, Wang XZ, Zhao X, Zhao W, Zhou TN, Zhang L. Optimal strategy of switching from clopidogrel to ticagrelor in Chinese acute coronary syndrome patients with complicated coronary artery disease: the switching from clopidogrel to ticagrelor (SHIFT-CACS) study. Chin Med J (Engl). 2019 Oct 5;132(19):2292-2299. doi: 10.1097/CM9.0000000000000444. PMID 31567375